CLINICAL TRIAL: NCT02067715
Title: Effectiveness of Sealed In-office Bleaching Technique: Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, André Luis Faria e Silva, Dr, Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFS001
Record Dates: First submitted 2014-02-15; First posted 2014-02-20 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Tooth Discoloration
Keywords: Tooth Discoloration; Bleaching Agents; Tooth Bleaching
MeSH Terms: conditions — Tooth Discoloration | interventions — Tooth Bleaching

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sealed bleaching Protocol (Experimental): The 35% hydrogen peroxide gel will be mixed and applied over the buccal surfaces of teeth. The bleaching agent will remain for 45-min application without replacement of peroxide. However, a customized tray will be placed over the bleaching agent during entire permanence of peroxide (45 minutes).
  Interventions: Drug: Tooth bleaching
- Conventional Bleaching Protocol (Active Comparator): The 35% hydrogen peroxide gel will be mixed and applied over the buccal surfaces of teeth. The bleaching agent will remain for 45-min application without replacement of peroxide.
  Interventions: Drug: Tooth bleaching

INTERVENTIONS:
Drug: Tooth bleaching — The bleaching agent will be used in a single-application of 45 minutes.
  Other Names: 35% hydrogen peroxide based bleaching agent, Whiteness HP Maxx, FGM, Joinville, SC, Brazil.

SUMMARY:
Thus, the aim of this study is to evaluate the sealed bleaching technique on tooth sensitivity and bleaching efficacy. The hypothesis is that the sealed bleaching technique reduce the tooth sensitivity when compared to conventional technique, without alters the bleaching efficacy.

DETAILED DESCRIPTION:
This is a randomized, single-blind, and controlled trial with a parallel group and an equal allocation rate to receive either one of two treatments, whereas the sealed technique is the experimental intervention and the conventional technique is control one.

PICO Question:

P (Population) - Patients of dentistry service of Federal University of Sergipe.

I: (Intervention) - In-office bleaching using 35% hydrogen peroxide bleaching agent covered with a customized tray.

C: (Control) - In-office bleaching using 35% hydrogen peroxide bleaching agent covered without a customized tray.

O: (Outcomes) - Primary outcomes: presence of tooth sensitivity during the bleaching procedure; Secondary outcome: Bleaching efficacy.

Sample Patients attempted in clinical service of Federal University of Sergipe requiring tooth bleaching will be recruited for this trial. For sample size calculation was considered 80% of test power, significance level of 5%, the presence of tooth sensitivity of 90% at control intervention and 40% at experimental intervention. These levels of sensitivity were based in pilot study. Thus the sample size for a proportions test (SigmaStat 3.5 (Systat Software, Point Richmond, USA) was 17 participants for each intervention.

Randomization Previously to beginning of study, a blocked randomisation list will be created using the website www.sealedenvelope.com, using block size of 4, by an operator different from those who will be perform the bleaching procedures. The bleaching protocol for each participant will be placed into a sealed envelope, while this only will be opened in the moment of bleaching procedure.

Evaluations During the permanence of bleaching agent, the tooth sensitivity will be monitored and the scores (VAS and verbal scale) will be recorded at 20th and 40th minute. The score also will be recorded immediately after the bleaching agent removal. In the after day, the participants will be argued (only verbal scale) about the maximum level of sensitivity during the first 24 hours after bleaching procedure and in 24th hour after this. A week after the bleaching procedure, the scores based on shade guides will be recorded again. For CIE L*a*b* measurement, ΔE will be calculated by the following equation: ∆E= [(∆L)2 + (∆a)2 + (∆b)2]1/2, while ∆L = L1 - L0; ∆a = a1 - a0; e ∆b = b1 - b0. After the shade evaluation, a new bleaching procedure, using the same protocol, will be performed in this second appointment and the same measurements of tooth sensitivity will be performed similarly to first one. After a week of second session, only the shade will be evaluated.

Blinding Once that it is not possible to blind the operators responsible by bleaching procedures and the participants, only the operators responsible by evaluations and by statistical analysis will be blinded.

Analysis of data The average of scores corresponding to shade guides will be calculated for each participant in the three moments of evaluation. Data will be submitted to Friedman and Man-Whitney tests. The average of ∆E will be calculated for each participant in the two moments of re-evaluation, while the data will be submitted to two-way ANOVA (protocol x moment of evaluation). Data for tooth sensitivity scores will be submitted to Friedman and Man-Whitney tests. The multiple-comparison test of Tukey will be used when necessary. The number of participants presenting any sensitivity during each session of bleaching will be calculated, while the percentage of these participants for each protocol will be calculated using Chi-square test. All statistical analysis will be performed with significant level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old patients of both genders presenting good general/oral health;
* All maxillary anterior teeth presenting shade equal or darker than 2M2 at Vita bleachguide guide (Vita-Zahnfabrik, Alemanha)
* Signed the form accepting to participate of this study.

Exclusion Criteria:

* Presence of caries lesions, restorations and/or endodontic treatment at any maxillary anterior teeth.
* Undergone tooth-whitening procedures;
* Pregnant/lactating;
* Smokers;
* Presence of periodontal diseases;
* Presence of severe tooth discoloration by tetracycline stains or fluorosis;
* Any kind of medicine, bruxism habits or any other pathology that can cause sensitivity (such as recession, dentin exposure);
* Continuous use of drugs with anti-inflammatory actions.
* Presence of tooth hypersensitivity at baseline measurement;
* Non-attendance to any session of evaluation or bleaching;

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Tooth sensitivity | During the bleaching procedure
  The tooth sensitivity will be assessed using a Visual analogue (VAS) and verbal scales. VAS consisted of a 10-cm color scale from green (no sensitivity) to red (unbearable sensitivity). A slightly air-stream will be applied over the buccal surfaces of the central incisors, and the patients will record their sensitivity perception by pointing with a pen on the scale. The distance between the marking and the border of scale, relative to the absence of sensitivity will be measured. The measurements will be scored according to: 0 - until 2-cm; 1 - between 2.1 and 4-cm; 2 - between 4.1 and 6-cm; 3 - between 6.1 and 8-cm; 4 - between 8.1 and 10-cm. For verbal scale, the patient will relate her/his level of sensitivity in a scale from 0 to 4, while 0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe. Participants presenting score different from 0 for any scale in this evaluation time will be excluded.

SECONDARY OUTCOMES:
Bleaching Effectiveness | Before the bleaching procedures and 7 days after this.
  The color evaluation will be performed using CIE L*a*b* color system, classical Vita guide and Vita bleachguide. For the CIE L*a*b* and classical vita guide, the shade will be determined using a spectrophotometer (Easy Shade Compact, Vita-Zahnfabrik, Bad Säckinge, Germany). The spectrophotometer also will inform the shade in classical Vita guide. The shades of this guide will be arranged in scores from highest (B1) to lowest (C4) values. Two calibrated examiners will evaluate the shade of teeth using the Vita Bleachguide. For calibration purposes, the teeth shades of five participants (whom will be did not include in the sample) will be evaluated individually by each examiner. A level of agreement higher than 80% must be reached before to begin the study evaluation. During the study, if disagreements arose, they will reach a consensus before dismissing the patient. For this guide, the shades also will be arranged in scores from highest (0M1) to lowest (5M3) values.

CONTACTS AND LOCATIONS:
Overall Officials: Andre L Faria-e-Silva, PhD, Study Chair — Universidade Federal de Sergipe
Locations (1):
- Universidade Federal de Sergipe, Aracaju, Sergipe, Brazil

REFERENCES:
- [Background] Reis A, Tay LY, Herrera DR, Kossatz S, Loguercio AD. Clinical effects of prolonged application time of an in-office bleaching gel. Oper Dent. 2011 Nov-Dec;36(6):590-6. doi: 10.2341/10-173-C. Epub 2011 Sep 13. PMID 21913864
- [Background] Kwon SR, Wertz PW, Dawson DV, Cobb DS, Denehy G. The relationship of hydrogen peroxide exposure protocol to bleaching efficacy. Oper Dent. 2013 Mar-Apr;38(2):177-85. doi: 10.2341/11-351-L. Epub 2012 Jul 7. PMID 22770431